CLINICAL TRIAL: NCT07209436
Title: Impact of Pectoral Versus Paravertebral Blocks on Pain and Physical Well-Being in Implant-Based Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Colwell (Other)
Responsible Party: Sponsor-Investigator, Amy Colwell, Sponsor-Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-544
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Reconstruction
Keywords: Breast Reconstruction; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral Block (Active Comparator): Paravertebral block at preop
  Interventions: Procedure: Paravertebral block (single injection)
- Pectoral Block (Experimental): Pectoral block at preop
  Interventions: Procedure: Pectoral block

INTERVENTIONS:
Procedure: Paravertebral block (single injection) — Paravertebral block at preop
  Arms: Paravertebral Block
Procedure: Pectoral block — Pectoral block at preop
  Arms: Pectoral Block

SUMMARY:
The broad aim of this study is to compare the effectiveness of paravertebral and pectoral blocks on pain and physical well-being of patients undergoing immediate implant-based breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years or older
* Scheduled for unilateral or bilateral immediate implant-based breast reconstruction
* Therapeutic or prophylactic indication
* Patient understands the study procedures and objectives and is willing to participate
* Patient willing to and capable of providing informed consent

Exclusion Criteria:

* Delayed breast reconstruction
* Allergy or contraindication to local anesthetics (PVB or PECS blocks)
* History of radiation therapy
* Planned sedation or general anesthesia protocol variation
* Morbid obesity as defined as a BMI greater than 40 kg/m2
* Renal insufficiency
* Chronic pain syndrome or central sensitization disorders (e.g., fibromyalgia, CRPS)
* Use of implanted pain devices or neuromodulators
* Pre-existing neurological deficits in the surgical field
* Current chronic opioid use (daily use within the 2 weeks before surgery and duration of use greater than 4 weeks)
* Use of any nerve medications in the past 6 months, including antiepileptic medications (gabapentin, carbamazepine)
* History of drug or alcohol abuse or habitual alcohol intake greater than two standard drinks per day (e.g., two beers, two glasses of wine, or two mixed drinks)
* Any comorbidity that results in moderate or severe functional limitation, inability to communicate with the investigators or hospital staff
* History of a psychiatric disorder which would interfere with the study procedure
* Incarceration
* Any issue that at the discretion of the investigator would contraindicate the subject's participation
* Inability to understand the procedures and objectives of the study
* Inability to or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Patient-reported physical well-being and breast symptoms | 12 Months
  Patient-reported physical well-being and breast symptoms will be evaluated using the Breast Quality of Life Physical Well-Being and Breast Symptoms scales. Values are scores from 0 to 100, with higher scores indicating better satisfaction or quality of life for patients undergoing breast surgery, such as those with breast cancer. These scores are derived from patient-reported outcome measures across different domains like satisfaction with breasts, psychosocial well-being, physical well-being (chest and abdomen), and sexual well-being.
Brief Pain Inventory (BPI) Scoring | 12 Months
  The BPI is a self-report questionnaire that assesses pain intensity and interference. It consists of two parts:
  Pain Severity: Measures the intensity of pain using a 0-10 scale, where 0 is "no pain" and 10 is "worst possible pain." Pain Interference: Measures how much pain interferes with daily activities using a 0-10 scale for seven items (e.g., general activity, mood, sleep).
  Calculation of Scores:
  Pain Severity Score: Add up the scores for the four pain severity questions (worst pain, least pain, average pain, current pain) and divide by 4.
  Pain Interference Score: Add up the scores for the seven pain interference questions and divide by 7.
  Interpretation:
  Pain Severity:
  0-3: Mild pain 4-6: Moderate pain 7-10: Severe pain
  Pain Interference:
  Higher scores indicate greater interference with daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Colwell, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No